CLINICAL TRIAL: NCT01883141
Title: Left Ventricular MultiSpot Pacing for CRT (iSPOT)
Acronym: iSPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iSPOT
Record Dates: First submitted 2013-05-24; First posted 2013-06-21 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrophysiological Study (Experimental): Subjects will receive pacing from one right ventricular lead and one left ventricular catheter/lead with multiple LV pacing spots during electrophysiological study procedure
  Interventions: Procedure: Electrophysiological Study

INTERVENTIONS:
Procedure: Electrophysiological Study — Subjects will receive pacing from one right ventricular lead and one left ventricular catheter/lead with multiple LV pacing spots

SUMMARY:
The purpose of the iSPOT Study is to evaluate the contractility using positive left ventricular (LV) dP/dt max across LV pacing site(s) in patients indicated for cardiac resynchronization therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for cardiac CRT or CRT-D device according to current applicable European Society of Cardiology (ESC)/American Heart Association (AHA) guidelines
* Subject has a left bundle branch block (LBBB) conduction pattern
* Subject is in stable sinus rhythm at the time of implant (no atrial arrhythmias lasting > 30 seconds during the last 2 weeks prior to inclusion and no documented atrial fibrillation (AF) episodes allowed during the last 2 weeks prior to inclusion)
* Subject receives optimal heart failure oral medical therapy (ACE inhibitor and/or angiotensin receptor blockers (ARB) and Beta Blockers), and is on a stable medication scheme for at least 1 month prior to enrollment
* Subject (or the legal guardian) is willing to sign informed consent form
* Subject is 18 years or older or as specified minimal age per local law/regulation

Exclusion Criteria:

* Subject has permanent atrial fibrillation/ flutter or tachycardia
* Subject experienced recent myocardial infarction (MI), within 40 days prior to enrollment
* Subject underwent coronary artery bypass graft (CABG) or valve surgery, within 90 days prior to enrollment
* Subject is post heart transplantation, or is actively listed on the transplantation list
* Subject is implanted with a left ventricular assist device (LVAD)
* Subject is on chronic renal dialysis
* Subject has severe renal disease (defined as estimated Glomerular Filtration Rate (equation provided by Modification of Diet in Renal Disease study): (eGFR) < 30 mL/min/1.73m2)
* Subject is on continuous or uninterrupted infusion (inotropic) therapy for heart failure (≥ 2 stable infusions per week)
* Subject has severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated within study period)
* Subject has complex and uncorrected congenital heart disease
* Subject has a mechanical heart valve
* Pregnant or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth control
* Subject is enrolled in one or more concurrent studies that would confound the results of this study
* Subject is already implanted with a device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Sterlinski, Dr., Principal Investigator — Warsaw Hospital
Locations (8):
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis Aalst, Aalst
  - Universitair Ziekenhuis Gent, Ghent
- Barzilai Medical Center, Ashkelon, Israel
- Poland (3):
  - Klinika Choroby Wieńcowej, Warsaw
  - Klinika Zaburzeń Rytmu Serca, Warsaw
  - Medical University of Silesia, Zabrze
- United Kingdom (2):
  - Guys and St. Thomas NHS Trust, London
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Jackson T, Lenarczyk R, Sterlinski M, Sokal A, Francis D, Whinnett Z, Van Heuverswyn F, Vanderheyden M, Heynens J, Stegemann B, Cornelussen R, Rinaldi CA. Left ventricular scar and the acute hemodynamic effects of multivein and multipolar pacing in cardiac resynchronization. Int J Cardiol Heart Vasc. 2018 Apr 10;19:14-19. doi: 10.1016/j.ijcha.2018.03.006. eCollection 2018 Jun. PMID 29946558

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled Patients: Patients who signed informed consent
Period: Overall Study
Arm/Group | Enrolled Patients
Started | 31
Passing Eligibility (Passing inclusion and exlcusion criteria) | 30
EP Study Performed | 30
Usable EP Data (Electrical instability (N=1), Technical failure (N=2), No veins available for lead placement (N=1)) | 26
BiV Pacing-Distal | 24
BiV Pacing-Mid | 25
BiV Pacing-Standard Therapy (Proximal pacing) | 26
Multispot-pacing | 24
BiV Pacing-Anterior | 23
Biv Pacing-Posterior | 22
Multivein | 23
Completed | 31 (Exit form with exit reason available)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Eligible Patients: The study enrolled 31 patients of which 30 patients fulfilled the inclusion and exclusion criteria.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Number; unit: participants]
  Belgium | 6
  Poland | 20
  United Kingdom | 3
  Israel | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Positive Left Ventricular (LV) dP/dt Max (mm HG/Sec) of Multispot LV Pacing Configuration Compared to Normal Biventricular Pacing
Description: Measure the percentage change in positive left ventricular (LV) dP/dt max (mm HG/sec) of multispot LV pacing configuration compared to normal biventricular pacing in patients undergoing a research study, an electrophysiological exploratory procedure or cardiac resynchronization therapy (CRT) implant. The percentage changes correspond to a percentage change between a pacing configuration (pacing on, e.g., Multispot pacing) and baseline (LV pacing off). There are several repetitions of pacing off and on for each pacing configuration. For one repetition, the percentage change is determined as ([median dP/dt max during pacing On] - (median baseline dP/dt max during pacing Off])/[median dP/dt max during pacing Off]. From all percentage changes for a given pacing configuration and subject, a regression analysis is performed to determine the regression predicted highest percentage change. The presented percentage change is the average over all subjects.
Time Frame: Participants will be followed for the time of the EP procedure, which has an average duration of 2 to 3 hours
Population: Patients underwent an electrophysiological (EP) visit during which multispot, multivein and biventricular (BiV) pacing was performed for each patient. From the 30 eligible patients, 4 patients were excluded from analysis (EP data collection issues: n = 4).
Measure: Mean (Standard Error); unit: percentage change LV dP/dt max
Arm/Group | Eligible Patients
Number analyzed (Participants) | 26
percentage change LV dP/dt max
  BiV distal: number analyzed (Participants) | 24
  BiV distal | 28.38 (3.15)
  BiV mid: number analyzed (Participants) | 25
  BiV mid | 28.58 (2.62)
  BiV proximal | 30.05 (2.75)
  Multispot: number analyzed (Participants) | 24
  Multispot | 31.04 (3.25)
  BiV anterior: number analyzed (Participants) | 23
  BiV anterior | 22.17 (2.31)
  BiV posterior: number analyzed (Participants) | 22
  BiV posterior | 30.05 (3.7)

2. Secondary Outcome: Percentage Change in Positive Left Ventricular (LV) dP/dt Max (mm HG/Sec) of Multi-vein LV Pacing Configuration Compared to Normal Biventricular Pacing
Description: Measure the percentage change in positive left ventricular (LV) dP/dt max (mm HG/sec) of multi-vein LV pacing configuration compared to normal biventricular pacing in patients undergoing a research study, an electrophysiological exploratory procedure or CRT-implant. The percentage changes correspond to a percentage change between a pacing configuration (pacing on, e.g., Multispot pacing) and baseline (LV pacing off). There are several repetitions of pacing off and on for each pacing configuration. For one repetition, the percentage change is determined as ([median dP/dt max during pacing On] - (median baseline dP/dt max during pacing Off])/[median dP/dt max during pacing Off]. From all percentage changes for a given pacing configuration and subject, a regression analysis is performed to determine the regression predicted highest percentage change. The presented percentage change is the average over all subjects.
Time Frame: Participants will be followed for the time of the EP procedure, which has an average duration of 2 to 3 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage change LV dP/dt max
Arm/Group | Eligible Patients
Number analyzed (Participants) | 26
percentage change LV dP/dt max
  BiV distal: number analyzed (Participants) | 24
  BiV distal | 28.38 (3.15)
  BiV mid: number analyzed (Participants) | 25
  BiV mid | 28.58 (2.62)
  BiV proximal | 30.05 (2.75)
  BiV anterior: number analyzed (Participants) | 23
  BiV anterior | 22.17 (2.31)
  BiV posterior: number analyzed (Participants) | 22
  BiV posterior | 30.05 (3.7)
  Multivein: number analyzed (Participants) | 23
  Multivein | 30.83 (3.44)

3. Secondary Outcome: Percentage Change in Positive Left Ventricular (LV) dP/dt Max (mm HG/Sec) of Multi-vein LV Pacing Configuration Compared to Multispot LV Pacing Configuration
Description: Measure the percentage change in positive left ventricular (LV) dP/dt max (mm HG/sec) of multi-vein LV pacing configuration compared to multispot LV pacing in patients undergoing a research study, an electrophysiological exploratory procedure or CRT-implant. The percentage changes correspond to a percentage change between a pacing configuration (pacing on, e.g., Multispot pacing) and baseline (LV pacing off). There are several repetitions of pacing off and on for each pacing configuration. For one repetition, the percentage change is determined as ([median dP/dt max during pacing On] - (median baseline dP/dt max during pacing Off])/[median dP/dt max during pacing Off]. From all percentage changes for a given pacing configuration and subject, a regression analysis is performed to determine the regression predicted highest percentage change. The presented percentage change is the average over all subjects.
Time Frame: Participants will be followed for the time of the EP procedure, which has an average duration of 2 to 3 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage change LV dP/dt max
Arm/Group | Eligible Patients
Number analyzed (Participants) | 26
percentage change LV dP/dt max
  Multispot: number analyzed (Participants) | 24
  Multispot | 31.04 (3.25)
  Multivein: number analyzed (Participants) | 23
  Multivein | 30.83 (3.44)

4. Secondary Outcome: Correlation of Blood Pressure, Electrograms (EGMs) and Electrocardiographic Mapping Measurements With the Positive LV dP/dt Max Values
Description: Correlate blood pressure, EGMs and electrocardiographic mapping measurements with the percentage change LV dP/dt max values obtained during each of the three pacing configurations BiV (BiV distal, BiV mid, BiV proximal, BiV anterior, BiV posterior), MultiVein and MultiSpot. Correlation will be summarized over all pacing configurations and time points since the interest is in the overall correlation between LV dP/dt max and other measurements, not in the correlation per pacing configuration or per time point. A linear mixed effects models as described in Roy, Biometrical Journal 48 (2006) 2, 286- 301 was used for the diastolic and systolic blood pressures. Due to the convergence problems for the linear mixed for Q-LV and QRS, the general linear model as described in Blank & Altman, Biometrical Journal 310 (1995), p 446, was used for Q-LV and QRS.
Time Frame: Participants will be followed for the time of the EP procedure, which has an average duration of 2 to 3 hours
Population: Patients underwent an electrophysiological (EP) visit during which multispot, multivein and biventricular (BIV) pacing was performed for each patient. From the 30 eligible patients, 4 patients were excluded from analysis due to EP data collection issues.
Measure: Number; unit: Correlation coefficient
Arm/Group | Eligible Patients
Number analyzed (Participants) | 26
Correlation coefficient
  Systolic blood pressure (Codan System) | 0.63
  Diastolic blood pressure (Codan system) | 0.45
  Systolic blood pressure (Nexfin system) | 0.37
  Diastolic blood pressure (Nexfin system) | 0.23
  QRS duration ratio | -0.20
  Q-LV | 0.52

5. Secondary Outcome: Use of Non-invasive Measurements to Identify Pacing Configuration With Highest Positive LV dP/dt Max
Description: Evaluate whether the non-invasive measurements (Nexfin blood pressures) that are also collected during the study can identify the pacing configuration with the highest percentage change LV dP/dt max. For each patient and all time points of data collection, a regression analysis was applied to determine the highest predicted percentage change LV dP/dtmax or percentage change Nexfin pressure per configuration. The Kappa statistic was then determined based on a 7x7 contingency table where the rows and columns corresponded to the pacing configurations. There is no interest in determining the agreement statistics Kappa per time point or per configuration since the interest of this analysis is in the overall agreement between LV dP/dt max and non-invasive measurements.
Time Frame: Participants will be followed for the time of the EP procedure, which has an average duration of 2 to 3 hours
Population: From the 30 eligible patients, 4 patients were excluded from analysis due to EP data collection issues and 2 patients were excluded since no blood pressure was collected non-invasively using a Nexfin system.
Measure: Number (95% Confidence Interval); unit: Kappa statistic
Arm/Group | Eligible Patients
Number analyzed (Participants) | 24
Kappa statistic
  Systolic blood pressure (Nexfin system) | 0.33 [0.09 to 0.58]
  Diastolic blood pressure (Nexfin system) | 0.33 [0.09 to 0.56]

6. Secondary Outcome: Within Patient Variability in Positive LV dP/dt Max
Description: Evaluate the within patient variability in positive LV dP/dt max measurements. The standard deviation of the percentage change LV dP/dt max between pacing configurations will be evaluated to obtain information for future sample size calculations for the primary outcome.The standard deviation is summarized over all available subjects and could be used as an estimate of within patient variability for future sample size calculations for the primary outcome.
Time Frame: Participants will be followed for the time of the EP procedure, which has an average duration of 2 to 3 hours
Population: as for outcome 4
Measure: Number; unit: percentage change
Arm/Group | Eligible Patients
Number analyzed (Participants) | 26
percentage change
  Multispot to BiV distal: number analyzed (Participants) | 23
  Multispot to BiV distal | 7.9
  MultiSpot to BiV proximal: number analyzed (Participants) | 24
  MultiSpot to BiV proximal | 5.6
  MultiSpot to BiV mid: number analyzed (Participants) | 24
  MultiSpot to BiV mid | 7.1
  MultiSpot to BiV anterior: number analyzed (Participants) | 21
  MultiSpot to BiV anterior | 11.0
  MultiSpot to BiV posterior: number analyzed (Participants) | 20
  MultiSpot to BiV posterior | 13.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to study exit. All types of adverse events (not only cardiovascular) were collected. Median number of days between enrollment and exit was 8 days with a minimum of 0 and a maximum of 116 days.
Arm/Group | Enrolled Patients
Serious Adverse Events (participants affected / at risk) | 5/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Patients (N=31)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Lead dislodgement (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less